CLINICAL TRIAL: NCT05285397
Title: Liraglutide's Effect on Weight Loss in Patients After Secondary Bariatric Surgery ; a Randomized Double-blind Controlled Study.
Brief Title: Effect of Liraglutide on Weight Loss in Patients Who Have Undergone Revisional Bariatric Surgeries.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Ass. Prof. of General surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Liraglutide1
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Morbid Obesity
Keywords: Liraglutide; Morbid obesity; secondary bariatric surgery; revisional bariatric surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide (Experimental): drug starts 6 weeks post-operative until 6 months SC injection dose starting 0.6 mg/day and weekly up titrated until 3.0 mg/day
  Interventions: Drug: Liraglutide Pen Injector [Saxenda]
- Control (No Intervention): Patients with no weight loss drug intervention after bariatric surgery

INTERVENTIONS:
Drug: Liraglutide Pen Injector [Saxenda] — Subcutaneous injection of GLP-1 agonist
  Arms: Liraglutide

SUMMARY:
Our primary objective is to assess the effect of Liraglutide on weight loss in patients who have undergone secondary bariatric surgeries. We set out to assess if Liraglutide is a viable option to augment weight loss in said category.

ELIGIBILITY:
Inclusion Criteria:

* Undergone primary bariatric surgery
* Need secondary bariatric surgery due to either weight regain (regained weight to have BMI > 35) or medical associated diseases

Exclusion Criteria:

* Prior use of GLP-1 agonist
* Past history of pancreatitis
* Personal or family history of medullary thyroid cancer
* Pregnancy or lactation
* Acute coronary syndrome
* Hepatic or renal dysfunction
* Active malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Percentage Total weight loss | 6 months
Percentage Excess body weight loss | 6 months

SECONDARY OUTCOMES:
Comorbidities | 6 months
Weight | 6 months
BMI | 6 months
HbA1C | 6 months
Fasting Blood Glucose (FBG) | 6 months
HOMA-IR | 6 months
Resolution of type 2 Diabetes Mellitus | 6 months
Blood pressure | 6 months
Lipid profile | 6 months
Sleep apnea | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Madina Women's Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thakur U, Bhansali A, Gupta R, Rastogi A. Liraglutide Augments Weight Loss After Laparoscopic Sleeve Gastrectomy: a Randomised, Double-Blind, Placebo-Control Study. Obes Surg. 2021 Jan;31(1):84-92. doi: 10.1007/s11695-020-04850-4. Epub 2020 Jul 12. PMID 32656729